CLINICAL TRIAL: NCT02491905
Title: Phase 2 Study to Assess Safety and Efficacy of HL Tablet on Reducing Hepatic Fat in Non-alcoholic Fatty Liver Disease Patients
Brief Title: Safety and Efficacy of HL Tablet in Non-alcoholic Fatty Liver Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-HS-HP-09-1
Record Dates: First submitted 2015-06-24; First posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- low dose HL tablet (Experimental): HL tablet which contains 66.7mg of active compound by oral administration, twice daily in an hour after meal
  Interventions: Drug: HL tablet
- high dose HL tablet (Experimental): HL tablet which contains 200mg of active compound by oral administration, twice daily in an hour after meal
  Interventions: Drug: HL tablet
- placebo group (Placebo Comparator): Placebo by oral administration, twice daily in an hour after meal
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HL tablet
  Arms: high dose HL tablet; low dose HL tablet
Drug: Placebo
  Arms: placebo group

SUMMARY:
This study evaluates the safety and efficacy of HL tablet on reducing hepatic fat in non-alcoholic fatty liver disease patients. The patients are allocated to three groups; low dose, high dose, and placebo control group.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 19 and 75
2. Non-alcoholic fatty liver disease patient

   * Diagnosed by abdomen ultrasonic examination
   * Non-drinker (alcohol intake per week : female-under 140g, male-under 210g)
3. ALT or AST higher than normal range (not over 4 times normal range)
4. Voluntary agreement and enrollment

Exclusion Criteria:

1. The ratio of AST/ALT over 2
2. Type I diabetes mellitus patient
3. Any dysfunction of liver besides non-alcoholic fatty liver disease
4. Alcoholic fatty liver disease patient or heavy drinker
5. Prior treatment with any medicine which affects the treatment of non-alcoholic fatty liver disease within 3 months
6. Patient taking any product which affects the BMI or hyperlipidemia
7. Any dyscrasia that investigator considers not to appropriate for this study
8. Bariatric surgery within 6 months
9. Any disease which is able to change the distribution of cytokines
10. Any treatment that affects liver functions within 1 month
11. Participation in other clinical trials within 3 months
12. Person who can not use MRS
13. Pregnancy or breast-feeding
14. Fertile women who do not use contraception
15. Sensitive to the investigational product
16. Any conditions that the investigator considers not to appropriate for this study

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
To assess the change of hepatic fat by Magnetic Resonance spectroscopy (MRS) after administration of HL tablet compared with baseline | 12 weeks

SECONDARY OUTCOMES:
Changes in Alanine Transaminase (ALT) | 8 and 12 week
Changes in Asparate Transaminase (AST) | 8 and 12 week
Changes in cholesterol | 8 and 12 week
Changes in triglyceride | 8 and 12 week
Changes in free fatty acid | 8 and 12 week
Changes in insulin resistance | 8 and 12 week
Changes in Body Mass Index (BMI) | 8 and 12 week

CONTACTS AND LOCATIONS:
Locations (1):
- Huons, Ansan, Kyeonggi-do, South Korea